CLINICAL TRIAL: NCT04621760
Title: Offering Women PrEP With Education and Shared Decision-making
Brief Title: The OPENS Trial: Offering Women PrEP (Aim 1)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Florida Department of Health (Other Government); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-014-FDOH; 3R01MD013565 (NIH)
Record Dates: First submitted 2020-10-09; First posted 2020-11-09 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-04

CONDITIONS: Human Immunodeficiency Virus Transmission; Sexually Transmitted Diseases
Keywords: Pre-exposure prophylaxis (PrEP); HIV prevention behaviors; HIV prevention methods; HIV education; African American, Latina, women of color; Shared decision making; Decision making, shared; Patient decision support; Patient decision aid
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: HIV Prevention Decision Support Tool (DST) - An interactive, tablet-based decision support tool that is designed to help women consider options to reduce their risk of HIV, with emphasis on PrEP as an emerging HIV prevention tool for women.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV Prevention DST Intervention (Experimental): Participants in this arm will receive the HIV prevention DST intervention and will receive the intervention immediately before their provider visit.
  Interventions: Behavioral: HIV Prevention Decision Support Tool (DST)
- Standard Counseling (Active Comparator): Participants in this arm will receive usual care.
  Interventions: Behavioral: Standard Counseling

INTERVENTIONS:
Behavioral: HIV Prevention Decision Support Tool (DST) — The tool is founded on principles of decision-science and developed in a systematic manner including pilot testing. The tool will present HIV prevention information through a tablet in the clinical setting. The decision support tool will address barriers to PrEP delivery, including 1) limited client knowledge about PrEP, 2) limited time to educate patients in busy clinics, 3) women's lack of knowledge of their own HIV vulnerability, and 4) hesitancy of women to initiate discussions about PrEP with providers due to judgmental attitudes and stigma. Also, the tool emphasizes the highly variable and individual nature of baseline risk.
  Arms: HIV Prevention DST Intervention
Behavioral: Standard Counseling — Participants in this arm will receive usual care.
  Arms: Standard Counseling

SUMMARY:
To address the significant barriers to PrEP implementation for those who were assigned female at birth and self-identify as a woman and address racial inequities in HIV prevention in the United States (US), a novel approach that accounts for multilevel influences is necessary. This study is one part of a multi-component project and involves a patient-level intervention in one public health family planning clinic in Duval County Florida, where the majority of patients are women of color. The area has one of the highest HIV incidence rates among women in the US. The investigators developed a tablet-based decision support tool that helps users learn about HIV vulnerabilities and HIV prevention strategies to inform how they consider options for reducing their likelihood of acquiring HIV. Participants will be randomized to use the HIV decision support tool before their visit or standard counseling (without the use of the tool) and will be surveyed about the use of the tool, experiences with HIV prevention counseling, and intentions about the use of HIV prevention. A subset of participants, all individuals who self-identify as a woman and as Black or Latina, will also complete a post-clinic visit interview. The investigators will follow-up with participants at three months following their initial visit to see if they have initiated the HIV prevention method(s) they chose at their visit. The main outcomes will include a quantitative and qualitative assessment of PrEP or other HIV prevention use, decisional certainty, and satisfaction with information about HIV prevention options.

Hypotheses:

1. Women who use the HIV prevention decision support tool will be more likely to have initiated PrEP within 3 months compared to women who received standard counseling at the time of their initial appointment.
2. The HIV prevention decision support tool will increase women's knowledge of PrEP and other HIV prevention methods compared to women who received standard counseling at the time of their initial appointment.
3. The HIV prevention decision support tool will increase participants' decisional certainty in their choice of an HIV prevention method compared to women who received standard counseling at the time of their initial appointment.

DETAILED DESCRIPTION:
Although 13% of the U.S. female population is Black, 60% of new HIV diagnoses in U.S. women occur among Black women. The South is the epicenter of the U.S. HIV epidemic, including in women, and Black Southern women are disproportionately affected: Black women account for 69% of new HIV diagnoses in women in the South. As the first highly effective, discrete, woman-controlled HIV prevention method, oral pre-exposure prophylaxis (PrEP) with tenofovir disoproxil fumarate/emtricitabine radically expands HIV prevention options for women. However, uptake of PrEP in U.S. women has lagged, particularly among groups most affected by HIV.

PrEP cascades outline the necessary steps for accessing PrEP, including screening and identifying eligible individuals, linkage to care, prescription, and initiation of PrEP. Data suggest there are multilevel barriers related to the process of screening for HIV risk in women and identifying potential PrEP candidates that may drive a significant drop off early in the PrEP cascade for women. Women report feeling judged by risk assessment questions and experience stigma around disclosing sexual practices. As a result, if screening is required to educate patients about PrEP - as is true in most clinical settings - many women for whom PrEP is appropriate may never learn about PrEP. Further, women have low levels of knowledge about HIV risk and HIV prevention options, and therefore will not seek out PrEP services themselves. By offering education to all women about vulnerabilities to HIV as well as information about HIV prevention methods including PrEP, at-risk women can circumvent these multifactorial barriers and request PrEP. Electronic decision support tools (DST), which have been used with success in a range of healthcare contexts including contraception, provide an efficient and private mechanism for this information-sharing step.

The study team developed a tablet-based tool that is designed to provide universal PrEP education and facilitate women's agency to identify their own risks and interest in PrEP. It was refined with iterative feedback from patient and community stakeholders and finalized based on cognitive testing.

The DST provides information about vulnerabilities to HIV and core characteristics of different HIV prevention methods, and then the opportunity to explore these characteristics in depth, including efficacy, safety and side effects. The user chooses the level of information that they wish to receive through the interactive interface, allowing for an individualized experience. Upon reaching the end of the tool, information on the tablet suggests that women ask their provider about HIV prevention methods they are interested in using, based on their preferences for method characteristics, and their questions in order to facilitate deliberation with the provider. The DST takes approximately 10 minutes to complete.

Approximately 200 women presenting to one reproductive health clinic in Duval County, Florida, will be randomized to standard counseling plus use of an HIV prevention DST, providing education about PrEP and encouraging self-assessment of HIV risk, or standard counseling alone. In addition to the experimental intervention, a subset of 40 participants (20 per arm) will be asked to allow audio-recording of their counseling sessions with a provider. A subset of up to 40 additional participants (20 per arm), all of whom self-identify as women of color, will be invited to complete one-hour, semi-structured interviews after their clinic visit about their experiences of using the DST, HIV prevention counseling, and decision making about PrEP.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as a woman (regardless of pregnancy status)
* Age 18 - 45 years
* Not known to be living with HIV (based on self-report)
* English-speaking
* Interested in participating

Exclusion Criteria:

* Unable to consent
* Currently using PrEP
* Those who were assigned male at birth and self-identify as a man
* Unwilling to be contacted in 3 months
* Already participated in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants have to identify as a woman.
Enrollment: 189 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Dehlendorf, MD, Principal Investigator — University of California, San Francisco; Akilah Pope, MD, Principal Investigator — Florida Department of Health in Duval County
Locations (1):
- Florida Department of Health in Duval County, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals will be handed a flyer about the study and eligibility criteria when they present to the front desk for check in.
  Interested individuals are then brought back to a private clinic room for an eligibility screening. Eligible individuals will then be enrolled into the study and randomized to either the control or intervention.
Pre-assignment Details: 3 individuals did not meet inclusion criteria. 4 individuals did not want to participate after learning more about the study.
Period: Overall Study
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Started | 95 (Protocol deviation resulted in 9 participants randomized to control not using the DST. 1 instance of technological issues and 8 instances of clinic time flow constraints.) | 94 (Protocol deviation due to user error resulted in 4 participants not being randomized to control or intervention. Those 4 participants were defaulted to the control group.)
Completed | 92 | 90
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV Prevention DST Intervention | Standard Counseling | Total
Number analyzed (Participants) | 95 | 94 | 189
Age, Customized [Count of Participants; unit: Participants] — Age collected on range from: 18-24; 25-29; 30-34; 35-44
  Participants
    Age: 18-24 years old | 27 | 30 | 57
    Age: 25-29 years old | 19 | 18 | 37
    Age: 30-34 years old | 30 | 25 | 55
    Age: 35-44 years old | 15 | 16 | 31
    Age: Missing | 4 | 5 | 9
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender identification of participant.
  Participants
    Gender: Female | 93 | 91 | 184
    Gender: Gender non-conforming or non-binary | 0 | 2 | 2
    Gender: Missing | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race and ethnicity of of participant.
  Participants
    Race/Ethnicity: African American/Black | 71 | 72 | 143
    Race/Ethnicity: Asian | 1 | 0 | 1
    Race/Ethnicity: Mixed race or multiracial | 5 | 4 | 9
    Race/Ethnicity: Native American | 0 | 1 | 1
    Race/Ethnicity: Pacific Islander | 1 | 0 | 1
    Race/Ethnicity: White | 14 | 14 | 28
    Race/Ethnicity: Other | 1 | 2 | 3
    Race/Ethnicity: Missing | 2 | 1 | 3
Parental Education [Count of Participants; unit: Participants] — Highest educational level reached by participant's parent.
  Participants
    8th grade or less | 4 | 4 | 8
    Some high school | 12 | 23 | 35
    High school graduate | 47 | 32 | 79
    Some college | 18 | 23 | 41
    College graduate or greater | 12 | 11 | 23
    Missing | 2 | 1 | 3
Yearly Income [Count of Participants; unit: Participants] — Total yearly income of participant.
  Participants
    < $10,000 | 41 | 38 | 79
    $10,000-$19,999 | 24 | 24 | 48
    $20,000-$29,999 | 15 | 15 | 30
    $30,000-$39,999 | 5 | 10 | 15
    Over $40,000 | 8 | 6 | 14
    Missing | 2 | 1 | 3
Educational Attainment [Count of Participants; unit: Participants] — Highest educational level reached by participant.
  Participants
    8th grade or less | 3 | 1 | 4
    Still in high school | 2 | 1 | 3
    < high school diploma | 13 | 6 | 19
    High school graduate | 44 | 49 | 93
    Some college | 27 | 29 | 56
    4-yr college graduate or more | 4 | 7 | 11
    Missing | 2 | 1 | 3
Ethnicity [Count of Participants; unit: Participants] — The ethnicity of the participant as either Hispanic/Latine or not Hispanic/Latine
  Participants
    Hispanic/Latine | 13 | 11 | 24
    Not Hispanic/Latine | 80 | 82 | 162
    Missing | 2 | 1 | 3
Housing Status [Count of Participants; unit: Participants] — Housing status of the participant.
  Participants
    Rent or own | 72 | 67 | 139
    Housing insecure | 21 | 26 | 47
    Missing | 2 | 1 | 3
Language Spoken at Home [Count of Participants; unit: Participants] — Language spoken in the participant's home.
  Participants
    English | 89 | 88 | 177
    Spanish | 1 | 0 | 1
    Mandarin | 1 | 0 | 1
    Other | 1 | 0 | 1
    Multiple | 1 | 5 | 6
    Missing | 2 | 1 | 3
Relationship Status [Count of Participants; unit: Participants] — The current relationship status of the participant.
  Participants
    Not in a relationship | 23 | 34 | 57
    In a relationship with one person | 66 | 54 | 120
    In a relationship with more than one person | 3 | 2 | 5
    Missing | 3 | 4 | 7
Percentage of monogamous participants [Count of Participants; unit: Participants] — Question finding out if the participant is monogamous, meaning in a relationship with only one other person.
  Participants | 62 | 53 | 115
Percentage of participants who had condomless vaginal sex, past 6 months [Count of Participants; unit: Participants] — A question finding out if the participant has had vaginal sex without a condom in the past 6 months.
  Participants | 64 | 61 | 125
Percentage of participants who had anal sex, past 6 months [Count of Participants; unit: Participants] — A question asking if the participant has had anal sex in the past 6 months.
  Participants | 8 | 7 | 15
STD Diagnosis History [Count of Participants; unit: Participants] — A question asking if the participant has ever been diagnosed with chlamydia, gonorrhea, hepatitis C, syphilis, or trichomonas.
  Participants
    Ever Had Chlamydia | 21 | 34 | 55
    Ever Had Gonorrhea | 11 | 14 | 25
    Ever Had Hepatitis C | 1 | 1 | 2
    Ever Had Syphilis | 0 | 2 | 2
    Ever Had Trichomonas | 14 | 18 | 32
Percentage of participants who have experienced domestic violence, ever [Count of Participants; unit: Participants] — A question asking if the participant has ever felt unsafe in a relationship.
  Participants | 9 | 7 | 16
Percentage of participants who engaged in binge drinking weekly or more frequently, past 6 months [Count of Participants; unit: Participants] — A question asking if the participant has engaged in binge drinking weekly or more frequently in the past 6 months.
  Participants | 6 | 9 | 15
Percentage of participants who have injected drugs, ever [Count of Participants; unit: Participants] — A question asking if the participant has ever injected drugs.
  Participants | 1 | 3 | 4
Percentage of participants who have used illicit substances, ever [Count of Participants; unit: Participants] — A question asking if the participant has ever used any illicit substance.
  Participants | 1 | 6 | 7
Percentage of participants who have experienced hunger, past year [Count of Participants; unit: Participants] — A question asking if the participant has gone hungry in the past year.
  Participants | 11 | 10 | 21
Percentage of participants who have been to jail or prison, ever [Count of Participants; unit: Participants] — A question asking if the participant has ever been to jail or prison.
  Participants | 17 | 23 | 40
Birth History [Count of Participants; unit: Participants] — A question asking how many times the participant has given birth.
  Participants
    Never | 16 | 24 | 40
    Once | 19 | 16 | 35
    Twice | 22 | 20 | 42
    Three or more times | 35 | 30 | 65
    Missing | 3 | 4 | 7
Percentage of participants who are currently breastfeeding [Count of Participants; unit: Participants] — A question asking if the participant is currently breastfeeding.
  Participants | 2 | 5 | 7
Percentage of participants who are currently pregnant [Count of Participants; unit: Participants] — A question asking if the participant is currently pregnant.
  Participants | 4 | 13 | 17
Percentage of participants who are currently trying to get pregnant [Count of Participants; unit: Participants] — A question asking if the participant is currently trying to get pregnant.
  Participants | 5 | 3 | 8
Percentage of participants who are currently using or plan to use condoms as contraception [Count of Participants; unit: Participants] — A question asking if the participant is using or planning to use condoms as a form of contraception.
  Participants | 36 | 34 | 70
Percentage of participants who are using or plan to use most/moderately effectively contraception [Count of Participants; unit: Participants] — A question asking if the participant is using or planning to use a mostly or moderately effective form of contraception.
  Participants | 70 | 60 | 130

OUTCOME MEASURES:

1. Primary Outcome: PrEP Prescriptions (As Measured by Chart Review)
Description: The number of participants who received a PrEP prescription within 3 months of their baseline visit, obtained by chart extraction from the medical record. Outcome is dichotomous (Yes, received a PrEP prescription /No, did not receive a PrEP prescription).
Time Frame: 3 months post baseline visit
Population: All participants who completed study activities at T1
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 90
Participants | 1 | 0
Statistical Analysis 1: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Test type: Superiority; p = 0.51, Fisher Exact — a priori threshold for statistical significance: 0.05

2. Secondary Outcome: Number of Patients Reporting PrEP Use
Description: Patients will be contacted at follow-up and asked if they took PrEP in the past 3 months regardless of where it was obtained. Outcome is dichotomous ("yes", initiated PrEP within 3 months of initial visit or "no", did not initiate PrEP within 3 months of initial visit).
Time Frame: 3 months post baseline visit
Population: Participants who completed one-month follow up survey
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 57 | 58
Participants | 1 | 1
Statistical Analysis 1: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Test type: Superiority; p = 0.62, Fisher Exact — threshold for significance: 0.05; one sided Fisher's exct test, given small cell sizes

3. Secondary Outcome: Change in Patient-Perceived HIV Risk
Description: We will measure the change in HIV risk perception in the next 6 months from pre- to post-visit at baseline. Response options include 4-point scale: 1 ("Not at all worried") to 4 ("Extremely worried").
Time Frame: Baseline, pre-intervention compared to immediately post baseline visit
Population: Participants who completed post-visit survey.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 90
Participants
  No Change | 77 | 85
  Increased Worry | 9 | 3
  Decreased Worry | 6 | 2
Statistical Analysis 1: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Test type: Superiority; p = 0.207, Fisher Exact — a priori threshold for significance: 0.05; Fisher's exact test used due to small sample size

4. Secondary Outcome: Patient-Perceived HIV Risk
Description: Participants will be asked about how worried they are about getting HIV in the next 6 months. Response options include 4-point scale of 1 ("Not at all worried") to 4 ("Extremely worried").
Time Frame: Immediately post baseline visit
Population: Participants who completed baseline survey.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 90
Participants
  Extremely worried | 2 | 4
  Very worried | 4 | 1
  A little worried | 11 | 13
  Not at all worried | 75 | 72
Statistical Analysis 1: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Test type: Superiority; p = 0.496, Fisher Exact — a priori threshold for significance: 0.05; Fisher's exact test used due to small cell size

5. Secondary Outcome: PrEP Knowledge
Description: Proportion of participants selecting the correct response to knowledge questions. Response options for each item are different. Higher score represents greater knowledge.
Time Frame: Immediately post baseline visit
Population: Participants who completed immediate post-visit survey
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 90
Participants
  PrEP is a daily pill to prevent HIV | 54 | 37
  PrEP is for all adults | 75 | 58
  PrEP will not work if taken once a week | 30 | 16
  PrEP does not prevent STDs other than HIV | 51 | 32
  PrEP side effects do not last forever | 51 | 23
  A baby could be born to HIV discordant parents without transmitting HIV | 46 | 31
  There is medication that you can take after sex to prevent HIV (PEP) | 51 | 21
  PrEP efficacy is > 95% | 43 | 49
Statistical Analysis 1: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Test comparing proportion correctly identifying "PrEP is a daily pill to prevent HIV"; Test type: Superiority; p = 0.02, Chi-squared — a priori threshold for significance: 0.05
Statistical Analysis 2: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Test comparing proportion correctly responding to prompt: "PrEP is for all adults"; Test type: Superiority; p = 0.01, Chi-squared — a priori threshold for significance: 0.05
Statistical Analysis 3: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Test comparing proportion who correctly identified: "PrEP will not work if taken once a week"; Test type: Superiority; p < 0.01, Chi-squared — a priori threshold for significance: 0.05
Statistical Analysis 4: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Test of proportion who correctly identified "PrEP does not prevent STDs other than HIV"; Test type: Superiority; p < 0.01, Chi-squared — a priori threshold for significance: 0.05
Statistical Analysis 5: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Test comparing proportion who correctly identified, "PrEP side effects do not last forever"; Test type: Superiority; p < 0.01, Chi-squared — a priori threshold for significance: 0.05
Statistical Analysis 6: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Test comparing proportion who correctly identified, "A baby could be norm to HIV discordant parents without transmitting HIV; Test type: Superiority; p = 0.03, Chi-squared — a priori threshold for significance: 0.05
Statistical Analysis 7: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Test comparing proportion who correctly identified "There is medication you can take after sex to prevent HIV"; Test type: Superiority; p < 0.01, Chi-squared — a priori threshold for significance: 0.05
Statistical Analysis 8: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Test for proportion who correctly identified "PrEP efficacy is > 95%"; Test type: Superiority; p = 0.29, Chi-squared — a priori threshold for significance: 0.05

6. Secondary Outcome: Decisional Conflict - Total Score
Description: Decisional Conflict scale: 16-item scale to measure decisional conflict. Response options range from 1-5 "strongly disagree" to "strongly agree". Items will be reverse-coded. Mean scores will be calculated, subtracted by 1, and multiplied by 25; scores range from 0 [no decisional conflict] to 100 [extremely high decisional conflict]. Higher scores represent high decisional conflict.
Time Frame: Immediately post baseline visit
Population: Participants who completed post-visit survey
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 90
units on a scale | 10 [0 to 25] | 0 [0 to 25]
Statistical Analysis 1: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Given strong positive skew of responses, transformed into a binary variable comparing those with lowest possible score versus higher score. Data then tested through tests of proportions; Test type: Superiority; p = 0.04, Chi-squared — a priori threshold for significance: 0.05

7. Secondary Outcome: Decisional Conflict - Uncertainty Subscore
Description: Three items from the Decisional Conflict scale will measure uncertainty: "I am clear about the best choice for me", "I feel sure about what to choose", and "the decision is easy for me to make". Response options range from 1-5 "strongly disagree" to "strongly agree". Items will be reverse-coded. Mean scores will be calculated, subtracted by 1, and multiplied by 25; scores range from 0 [feels extremely certain about best choice] to 100 [feels extremely uncertain about decision]. Higher scores represent greater decision uncertainty.
Time Frame: Immediately post baseline visit
Population: Participants who completed immediate post-visit survey
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 90
units on a scale | 16.7 [0 to 25] | 0 [0 to 25]
Statistical Analysis 1: Comparison: HIV Prevention DST Intervention vs Standard Counseling; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.02, Chi-squared — a priori threshold for significance: 0.05

8. Secondary Outcome: Decisional Conflict - Informed Subscore
Description: Three items from the Decisional Conflict scale will measure the informed subscale: "I know which options are available to me", "I know the benefits of each option", and "I know the risks and side effects of each option". Response options range from 1-5 "strongly disagree" to "strongly agree". Items will be reverse-coded. Mean scores will be calculated, subtracted by 1, and multiplied by 25; scores range from 0 [feels extremely informed] to 100 [feels extremely uninformed]. Higher scores represent a greater degree of feeling uninformed.
Time Frame: Immediately post baseline visit
Population: Participants who completed immediate post-visit survey
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 90
units on a scale | 0 [0 to 25] | 0 [0 to 25]
Statistical Analysis 1: Comparison: HIV Prevention DST Intervention vs Standard Counseling; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.05, Chi-squared — a priori threshold for significance: 0.05

9. Secondary Outcome: Decisional Conflict - Values Clarity Subscore
Description: Three items from the Decisional Conflict scale will measure values clarity: "I am clear about which benefits matter the most to me", "I am clear about which risks and side effects matter most to me", and "I am clear about which is more important to me (the benefits or the risks and side effects." Response options range from 1-5 "strongly disagree" to "strongly agree". Items will be reverse-coded. Mean scores will be calculated, subtracted by 1, and multiplied by 25; scores range from 0 [feels extremely clear about personal values for benefits and risks/side effects] to 100 [feels extremely unclear about personal values].
Time Frame: Immediately post baseline visit
Population: Participants who completed immediate post-visit survey
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 90
units on a scale | 12.5 [0 to 25] | 0 [0 to 25]
Statistical Analysis 1: Comparison: HIV Prevention DST Intervention vs Standard Counseling; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.03, Chi-squared — a priori threshold for significance: 0.05

10. Secondary Outcome: Decisional Conflict - Support Subscore
Description: Three items from the Decisional Conflict scale will measure support: "I have enough support from others to make a choice", "I am choosing without pressure from others", and "I have enough advice to make a choice". Response options range from 1-5 "strongly disagree" to "strongly agree". Items will be reverse-coded. Mean scores will be calculated, subtracted by 1, and multiplied by 25; scores range from 0 [feels extremely supported in decision making] to 100 [feels extremely unsupported in decision making].
Time Frame: Immediately post baseline visit
Population: Participants who completed immediate post-visit survey
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 90
units on a scale | 6.3 [0 to 25] | 0 [0 to 25]
Statistical Analysis 1: Comparison: HIV Prevention DST Intervention vs Standard Counseling; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.07, Chi-squared — a priori threshold for significance: 0.05

11. Secondary Outcome: Decisional Conflict - Effective Decision Subscore
Description: Four items from the Decisional Conflict scale will measure effective decision: "I feel I have made an informed choice", "my decision shows what is important to me", "I expect to stick with my decision", and "I am satisfied with my decision". Response options range from 1-5 strongly disagree to strongly agree. Items will be reverse-coded. Mean scores will be calculated, subtracted by 1, and multiplied by 25; scores range from 0 [good decision] to 100 [bad decision].
Time Frame: Immediately post baseline visit
Population: Participants who completed immediate post-visit survey
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 90
units on a scale | 16.7 [0 to 25] | 0 [0 to 25]
Statistical Analysis 1: Comparison: HIV Prevention DST Intervention vs Standard Counseling; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.10, Chi-squared — a priori threshold for significance: 0.05

12. Secondary Outcome: Interpersonal Quality of HIV Prevention Care
Description: Mean score of 4-item scale. Derived from the Person-Centered Contraceptive Care measure developed by the PI. Response options consist of 5-point Likert scale: 1 ("strongly disagree") to 5 ("strongly agree"). Scores will be dichotomized between 20 [excellent interpersonal quality of care] and less than 20 [poor interpersonal quality of care].
Time Frame: Immediately post baseline visit
Population: Participants who completed immediate post-visit survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 90
units on a scale | 17.2 (4.9) | 16.9 (5.3)
Statistical Analysis 1: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Given strong negative skew of responses, transformed into a binary variable comparing those with highest possible score versus higher score. Data then tested through tests of proportions; Test type: Superiority; p = 0.22, Chi-squared — a priori threshold for significance: 0.05

13. Secondary Outcome: Intention to Use Any HIV Prevention Method
Description: A one-time, one-item measure of plan to use HIV prevention method after the initial visit. Participants can select from "none", condoms, PrEP, post exposure prophylaxis (PEP), treatment as prevention, regular HIV testing (inclusive of partner), "still thinking about my options", or other method.
Time Frame: Immediately post baseline visit
Population: participants who completed immediate post-visit survey
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 90
Participants
  Any method | 88 | 87
  Abstinence | 38 | 39
  Condoms | 77 | 77
  PEP | 20 | 17
  PrEP | 19 | 15
  Regular HIV testing | 79 | 80
  Regular STD testing | 82 | 82
  Treatment as prevention | 58 | 66
Statistical Analysis 1: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Test type: Superiority; p = 0.51, Fisher Exact — a priori threshold for significance: 0.05; Fisher's exact test used due to small cell size

14. Secondary Outcome: Confidence in Decision to Use an HIV Prevention Method
Description: A one-time, one-item measure of certainty of plan to use HIV prevention after the initial visit. Participants can select from 4 options: 1 ("completely unsure"), 2 ("mostly unsure"), 3 ("mostly sure, but not 100%"), or 4 ("100% sure").
Time Frame: Immediately post baseline visit
Population: participants who completed immediate post-visit survey
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 90
Participants
  PrEP: number analyzed (Participants) | 19 | 15
  PrEP: I feel completely unsure | 2 | 2
  PrEP: I feel mostly unsure | 1 | 2
  PrEP: I feel mostly sure | 6 | 4
  PrEP: I feel 100% sure | 10 | 7
  Abstinence: number analyzed (Participants) | 38 | 39
  Abstinence: I feel completely unsure | 1 | 1
  Abstinence: I feel mostly unsure | 2 | 4
  Abstinence: I feel mostly sure | 9 | 6
  Abstinence: I feel 100% sure | 26 | 28
  Condoms: number analyzed (Participants) | 77 | 76
  Condoms: I feel completely unsure | 1 | 2
  Condoms: I feel mostly unsure | 0 | 3
  Condoms: I feel mostly sure | 18 | 12
  Condoms: I feel 100% sure | 58 | 59
  PEP: number analyzed (Participants) | 20 | 17
  PEP: I feel completely unsure | 1 | 3
  PEP: I feel mostly unsure | 1 | 1
  PEP: I feel mostly sure | 3 | 5
  PEP: I feel 100% sure | 15 | 8
  Regular HIV testing: number analyzed (Participants) | 79 | 80
  Regular HIV testing: I feel completely unsure | 0 | 3
  Regular HIV testing: I feel mostly unsure | 2 | 2
  Regular HIV testing: I feel mostly sure | 3 | 4
  Regular HIV testing: I feel 100% sure | 74 | 71
  Regular STD testing: number analyzed (Participants) | 82 | 82
  Regular STD testing: I feel completely unsure | 0 | 2
  Regular STD testing: I feel mostly unsure | 3 | 2
  Regular STD testing: I feel mostly sure | 7 | 3
  Regular STD testing: I feel 100% sure | 72 | 75
  Treatment as prevention: number analyzed (Participants) | 34 | 24
  Treatment as prevention: I feel completely unsure | 1 | 1
  Treatment as prevention: I feel mostly unsure | 1 | 4
  Treatment as prevention: I feel mostly sure | 4 | 0
  Treatment as prevention: I feel 100% sure | 28 | 19
Statistical Analysis 1: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Comparing confidence between treatment groups of those who said they intended to use PrEP; Test type: Superiority; p = 0.90, Fisher Exact — a priori threshold for significance: 0.05
Statistical Analysis 2: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Comparing confidence between treatment groups of those who said they intended to use abstinence; Test type: Superiority; p = 0.75, Fisher Exact — a priori threshold for significance: 0.05
Statistical Analysis 3: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Comparing confidence between treatment groups of those who said they intended to use PEP; Test type: Superiority; p = 0.32, Fisher Exact — a priori threshold for significance: 0.05
Statistical Analysis 4: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Comparing confidence between treatment groups of those who said they intended to use HIV testing; Test type: Superiority; p = 0.40, Fisher Exact — a priori threshold for significance: 0.05
Statistical Analysis 5: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Comparing confidence between treatment groups of those who said they intended to use STD testing; Test type: Superiority; p = 0.34, Fisher Exact — a priori threshold for significance: 0.05
Statistical Analysis 6: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Comparing confidence between treatment groups of those who said they intended to use Treatment as Prevention; Test type: Superiority; p = 0.10, Fisher Exact — a priori threshold for significance: 0.05

15. Secondary Outcome: Satisfaction With Information Received About HIV Prevention
Description: Participants will be asked a one-time question regarding satisfaction with HIV prevention counseling. Response options include: 1 ("I was not given any information about HIV), 2 ("very unsatisfied") 3 ("somewhat unsatisfied), 4 ("neither satisfied or unsatisfied"), 5 ("somewhat satisfied") and 6 ("very satisfied").
Time Frame: Immediately post baseline visit
Population: participants who completed immediate post-visit survey
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 90
Participants
  Very satisfied | 77 | 60
  Somewhat satisfied | 9 | 10
  Neither satisfied nor unsatisfied | 3 | 9
  Somewhat unsatisfied | 1 | 1
  Very unsatisfied | 2 | 1
  I was not given information about HIV prevention | 0 | 9
Statistical Analysis 1: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Test type: Superiority; p = 0.01, Chi-squared — a priori threshold for significance: 0.05

16. Secondary Outcome: Perceived Quality of Information Received About HIV Prevention
Description: Participants will be asked four questions about the perceived quality of the HIV prevention information patients received during their health care visit: 1) getting the information they needed, 2) the ease of understanding the information, 3) the trustworthiness of the information, and 4), the usefulness of the information. These questions will be asked of those who reported talking about HIV/HIV prevention during their visit with the healthcare provider or health educator OR those who talked to the healthcare provider or health educator about their chances of getting HIV. Response options are 1 to 5 "strongly disagree" to "strongly agree". Higher values indicate greater perceived quality.
Time Frame: Immediately post baseline visit
Population: participants who completed immediate post-visit survey
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 90
Participants
  I got all the information I needed (strongly agree) | 35 | 31
  Information was easy to understand (strongly agree) | 37 | 31
  Trusted the information given (strongly agree) | 35 | 32
  Found the information useful (strongly agree) | 33 | 31
Statistical Analysis 1: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Comparing proportions in response to prompt "The information was easy to understand"; Test type: Superiority; p = 0.26, Fisher Exact — a priori threshold for significance: 0.05
Statistical Analysis 2: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Comparing proportions in response to prompt: "I got all of the information I needed"; Test type: Superiority; p = 0.26, Fisher Exact — a priori threshold for significance: 0.05
Statistical Analysis 3: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Test type: Superiority; p = 0.59, Fisher Exact — a priori threshold for significance: 0.05
Statistical Analysis 4: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Comparing proportions in response to prompt: "The information felt useful to me"; Test type: Superiority; p = 0.17, Fisher Exact — a priori threshold for significance: 0.05

17. Secondary Outcome: Acceptability of HIV Prevention Methods
Description: Participants are asked to rate their preference for a method (even if they never used it). Participants can select from condoms, PrEP, PEP, partner HIV testing, regular STD testing, treatment as prevention or other method. The option, "never heard of it" is also included. Options for this scale range from 0 ("Terrible method for me") to 10 ("Great method for me").
Time Frame: Immediately post baseline visit
Population: participants who completed immediate post-visit survey
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 90
Participants
  Abstinence (great method for me) | 27 | 29
  Condoms (great method for me) | 35 | 40
  PEP (great method for me) | 18 | 14
  PrEP (great method for me) | 19 | 14
  HIV Testing (great method for me) | 48 | 48
  STD Tesating (great method for me) | 47 | 48
  Treatment as prevention (great method for me) | 24 | 20
Statistical Analysis 1: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Testing proportion of acceptability of abstinence method (proportion that responded "great for me"); Test type: Superiority; p = 0.74, Chi-squared
Statistical Analysis 2: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Testing proportion of acceptability of condoms method (proportion that responded "great for me"); Test type: Superiority; p = 0.59, Chi-squared
Statistical Analysis 3: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Testing proportion of acceptability of PEP method (proportion that responded "great for me"); Test type: Superiority; p = 0.66, Chi-squared
Statistical Analysis 4: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Testing proportion of acceptability of PrEP method (proportion that responded "great for me"); Test type: Superiority; p = 0.49, Chi-squared
Statistical Analysis 5: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Testing proportion of acceptability of HIV testing method (proportion that responded "great for me"); Test type: Superiority; p = 0.94, Chi-squared
Statistical Analysis 6: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Testing proportion of acceptability of STD testing method (proportion that responded "great for me"); Test type: Superiority; p = 0.95, Chi-squared
Statistical Analysis 7: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Testing proportion of acceptability of Treatment as prevention method (proportion that responded "great for me"); Test type: Superiority; p = 0.39, Chi-squared

18. Secondary Outcome: Acceptability of the Decision Support Tool
Description: Participants are asked four questions about their experiences using the DST (e.g., degree to which they got all the information they needed, found the information to be easy to understand, trust the information, and found information useful). Response items vary from strongly disagree to strongly agree.
Time Frame: Immediately post baseline visit
Population: group randomized to the DST
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 0
Participants
  Got all of the information I need from the DST (strongly agree or agree) | 82 | 0
  Information on the DST was easy to understand (strongly agree or agree) | 81 | 0
  I trusted the information on the DST (strongly agree or agree) | 83 | 0
  The information felt helpful to me (strongly agree or agree) | 71 | 0

19. Secondary Outcome: Perception of the Decision Support Tool
Description: Participants in the experimental arm will be asked about the degree to which they liked/disliked the tool. Response options vary: "I did not like it at all", "I somewhat disliked it", "I somewhat liked it", "I really liked it".
Time Frame: Immediately post baseline visit
Population: Group randomized to DST
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 0
Participants
  I really liked it: number analyzed (Participants) | 85 | 0
  I really liked it | 66 | 0
  I somewhat liked it | 18 |
  I somewhat disliked it | 1 |

20. Secondary Outcome: Satisfaction With the Decision Support Tool
Description: Participants in the experimental arm will be asked about the degree to which they were satisfied with the information in the tool. Response options vary from 1-5: "very unsatisfied" to "very satisfied".
Time Frame: Immediately post baseline visit
Population: Group randomized to the DST
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 0
Participants
  Very satisfied | 69 | 0
  Somewhat satisfied | 10 |
  Neither satisfied nor unsatisfied | 5 |
  Very unsatisfied | 1 |
  Missing | 7 |

21. Secondary Outcome: Recommend the Decision Support Tool
Description: Participants in the experimental arm will be asked whether they would recommend the tool a friend. Response options are "yes", "no", "unsure".
Time Frame: Immediately post baseline visit
Population: Group randomized to the DST
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 0
Participants | 81 | 0

22. Secondary Outcome: Willingness to Use the Decision Support Tool at Future Visits
Description: Participants in the experimental arm will be asked about whether they would use the tool again if they returned to the clinic. Response options are "yes", "no", "unsure".
Time Frame: Immediately post baseline visit
Population: Group randomized to the DST
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 92 | 0
Participants | 63 | 0

23. Secondary Outcome: HIV Prevention Method Use (Any Method - Planned or New Method)
Description: A self-reported measure of HIV prevention method use, including those who reported discontinuing the initial HIV prevention method(s) that were reported post-clinic visit. A response of "yes" to any of the following questions: since your [baseline] visit, have you used….for HIV prevention - abstinence, condoms, PEP, PrEP, regular HIV testing, treatment as prevention, regular sexually transmitted disease (STD) testing, other method. The outcome will be dichotomized to those who responded affirmatively vs other responses ("no"/"unsure").
Time Frame: 3 months post baseline visit
Population: participants who completed 3-month follow-up survey
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 57 | 58
Participants | 53 | 49
Statistical Analysis 1: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Test type: Superiority; p = 0.13, Fisher Exact — a priori threshold for significance: 0.05

24. Secondary Outcome: HIV Prevention Method Continuation
Description: A self-reported measure of HIV prevention method continuation. A response of "yes" to any of the following questions: are you still using - abstinence, condoms, PEP, PrEP, regular HIV testing, treatment as prevention, regular sexually transmitted disease (STD) testing, other method. The outcome will be dichotomized to those who responded "yes" vs "no".
Time Frame: 3 months post baseline visit
Population: participants who completed 3-month follow-up survey
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
Number analyzed (Participants) | 57 | 58
Participants | 53 | 48
Statistical Analysis 1: Comparison: HIV Prevention DST Intervention vs Standard Counseling; Test type: Superiority; p = 0.08, Fisher Exact — a priori threshold for significance: 0.05

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | HIV Prevention DST Intervention | Standard Counseling
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/94
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/94
Other Adverse Events (participants affected / at risk) | 0/95 | 0/94

LIMITATIONS AND CAVEATS:
COVID-19 disrupted normal clinic operations, including limiting HIV/PrEP counseling, and paused a state-wide PrEP campaign for cisgender women. This study was conducted at a single, publicly funded clinic with few providers and recruited primarily English-speaking participants and is not generalizeable to other populations. Further, there were too few participants who identified as non-cisgender women or reported injection drug use to report on experiences of those populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT04621760/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/60/NCT04621760/SAP_001.pdf
  • Informed Consent Form (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT04621760/ICF_002.pdf